CLINICAL TRIAL: NCT04399629
Title: Preschool Based Prevention Targeting Emotion Development in Young Children Facing Adversity
Brief Title: Trial of PCIT-ED in School for Preschoolers in Poverty
Acronym: PCIT-ED-ACES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: The Jennings School District (Unknown)
Responsible Party: Principal Investigator, Joan Luby, MD, Professor of Psychiatry, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 22-3250-18012
Record Dates: First submitted 2020-05-18; First posted 2020-05-22 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Childhood Mental Disorder
Keywords: Preschool; Parent-Child Relationship; Emotion Development; Therapy
MeSH Terms: conditions — Neurodevelopmental Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCIT-ED (Active Comparator): Parent-Child Interaction Therapy - Emotional Development (PCIT-ED) is a promising early intervention for depression that directly targets developing affective systems and builds on the empirical literature on emotion development and prevention.
  Interventions: Behavioral: PCIT-ED
- Parenting Wisely (Experimental): Online parenting training
  Interventions: Behavioral: Parenting Wisely

INTERVENTIONS:
Behavioral: PCIT-ED — 12 sessions of PCIT-ED therapy
  Arms: PCIT-ED
Behavioral: Parenting Wisely — Teaches parents how to set more effective limits
  Arms: Parenting Wisely

SUMMARY:
A shorted form of the previously tested, Parent Child Interaction Therapy Emotion Development (PCIT-ED) will be conducted with a sample of preschoolers who exhibit symptoms of behavioral problems as rated by teacher. Children aged 3-7 will be randomized to a 12-week PCIT-ED delivered by trained therapists in the school setting or an on-line parent training called "Parenting Wisely (PW)". Children will have a 60% chance of being randomized to PCIT-ED and 40% to PW. The treatment will be provided to eligible children in the Jennings School District at the school site. In order to test the efficacy of PCIT-ED, to estimate accurate effect sizes, and to investigate mediators and moderators of treatment response, participants will complete comprehensive pre- and post-assessments at Washington University School of Medicine Early Emotional Development Program.

Preschoolers over age 3 will be offered the option of enrolling in an add-on electroencephalography and magnetic resonance imagery study, to investigate neural changes associated with PCIT-ED or PW.

Compared to those randomized to PW, we expect preschoolers who undergo PCIT-ED will show significantly increased rates of remission of behavioral problems, greater reductions in symptoms, and decreases in impairment. We hypothesize that they will show significantly greater increases in emotional competence measured by the ability to accurately identify emotions in themselves and others and the ability to effectively regulate intense emotions. Compared to those on the PW, parents who undergo PCIT-ED will show significantly greater increases in emotion skill learning and reductions in MDD symptoms and parenting stress.

ELIGIBILITY:
Inclusion Criteria:

* Over the clinical threshold on the Teacher Report Form

Exclusion Criteria:

* Autism
* Major neurological disorder
* Participating in active weekly individual or family therapy

Ages: 48 Months to 83 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2019-09-26 (Actual); Primary Completion 2021-01-19 (Actual); Study Completion 2021-01-19 (Actual)

PRIMARY OUTCOMES:
McArthur Health and Behavior Questionnaire | completion of therapy (average of 12 weeks)
  The Health and Behavior Questionnaire was designed to assess children's mental health, physical health, and social and school functioning. The HBQ comprises multiple scales that measure children's symptoms (e.g., internalizing and externalizing symptoms and their subscales), physical health, social functioning (e.g., peer acceptance and rejection, prosocial behaviors), and school functioning (e.g., academic competence, school engagement). The HBQ also includes measures of children's health care utilization in the mental, physical, and school domains.
Teacher Report Form | completion of therapy (average of 12 weeks)
  This measure is used to obtain an overview of the child's behavior and functioning from the perspective of the teacher. The results of the form offer cross-informant comparisons in competencies, adaptive functioning and reported problems. This information is helpful for finding the child's strengths and where the child needs help.

SECONDARY OUTCOMES:
Eyberg Child Behavior Inventory | completion of therapy (average of 12 weeks)
  The Eyberg Child Behavior Inventory (ECBI) is a measure that asks parents to report on a list of thirty-six conduct problem behaviors in their child. It is designed for children ages 2-16 years. The ECBI includes an Intensity Scale, which measures the frequency of each problem behavior, and a Problem Scale, which reflects parents' tolerance of the behaviors and the distress caused. The ECBI is intended to assess both the type of behavior problems and the degree to which parents find them problematic.
Parent-Child Interaction: Marble Run and Drawing Task | completion of therapy (average of 12 weeks)
  The marble run task and the drawing task are observational measures of parent-child interactions used in preschool aged children. In the marble run task, parents and children are asked to build a marble run, replicating a picture of a marble run. The drawing task asks parents and children to together decide on something to draw on a blank sheet of paper and each contribute individual lines to the drawing, while sharing one marker. Both tasks were designed to elicit mild stress while also asking parents and children to work together. Both of these tasks (each lasting approximately three minutes) asks parents to help their child with the task but not complete it for them. Participants are videotaped while engaging in these tasks, and parents' behavior and emotions are coded.
Parenting Styles Questionnaire | completion of therapy (average of 12 weeks)
  The Parenting Style Questionnaire is an 81-item True/False measure that asks parents about their feelings regarding sadness, fear, and anger.
Parenting Styles and Dimensions Questionnaire | completion of therapy (average of 12 weeks)
  The PSDQ is a 62-item questionnaire that is designed to assess parenting style. The parent is given a list of 62 behaviors and asked how much they and their spouse exhibit each behavior.
Coping with Children's Negative Emotions Scale | completion of therapy (average of 12 weeks)
  The CCNES assesses how parents typically respond to their child's negative emotions. Parents are given 12 hypothetical situations in which their child is upset or angry. Each situation is accompanied with 6 possible ways to respond to the child, and the parent is asked to rate the likelihood that they will use each response.

CONTACTS AND LOCATIONS:
Overall Officials: Joan L Luby, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Early Emotional Development Program, St Louis, Missouri, United States

REFERENCES:
- [Background] Luby JL, Gilbert K, Whalen D, Tillman R, Barch DM. The Differential Contribution of the Components of Parent-Child Interaction Therapy Emotion Development for Treatment of Preschool Depression. J Am Acad Child Adolesc Psychiatry. 2020 Jul;59(7):868-879. doi: 10.1016/j.jaac.2019.07.937. Epub 2019 Jul 31. PMID 31376501
- [Background] Barch DM, Whalen D, Gilbert K, Kelly D, Kappenman ES, Hajcak G, Luby JL. Neural Indicators of Anhedonia: Predictors and Mechanisms of Treatment Change in a Randomized Clinical Trial in Early Childhood Depression. Biol Psychiatry. 2019 May 15;85(10):863-871. doi: 10.1016/j.biopsych.2018.11.021. Epub 2018 Dec 4. PMID 30583852 (Retraction: PMID 33153528 Biol Psychiatry. 2020 Dec 1;88(11):888)
- [Background] Luby JL, Barch DM, Whalen D, Tillman R, Freedland KE. A Randomized Controlled Trial of Parent-Child Psychotherapy Targeting Emotion Development for Early Childhood Depression. Am J Psychiatry. 2018 Nov 1;175(11):1102-1110. doi: 10.1176/appi.ajp.2018.18030321. Epub 2018 Jun 20. PMID 29921144
- [Derived] Hennefield L, Gilbert K, Donohue MR, Tillman R, McCoy A, Diggs G, Paul ZA, Kohl PL, Luby JL. Early Emotion Development Intervention Improves Mental Health Outcomes in Low-Income, High-Risk Community Children. Child Psychiatry Hum Dev. 2025 Oct;56(5):1457-1471. doi: 10.1007/s10578-023-01639-1. Epub 2024 Jan 14. PMID 38221601
- See also: Early Emotional Development Program Website — https://eedp.wustl.edu/